CLINICAL TRIAL: NCT00521248
Title: Buprenorphine for the Treatment of Neonatal Abstinence Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Steve Oversby, NIDA
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21DA018207-01 (NIH); R21DA018207-01 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2007-08-23; First posted 2007-08-27 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2009-12

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: Neonatal Abstinence Syndrome; buprenorphine; neonatal; opioid withdrawal
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral morphine solution (Active Comparator): Oral morphine solution
  Interventions: Drug: Oral morphine solution
- Buprenorphine (Experimental): Sublingual buprenorphine
  Interventions: Drug: buprenorphine

INTERVENTIONS:
Drug: buprenorphine — sublingual buprenorphine administered every 8 hours, titrated to control of abstinence symptoms
  Other Names: Buprenex (buprenorphine)
  Arms: Buprenorphine
Drug: Oral morphine solution — 0.4 mg/kg/day morphine every 4 hours
  Other Names: morphine
  Arms: Oral morphine solution

SUMMARY:
Neonatal abstinence syndrome is a disease that affects children who were exposed to opioid drugs prior to birth. Commonly used treatments at present include morphine or tincture of opium. Buprenorphine is a drug used in adults to treat narcotic dependence, but has not been used for Neonatal Abstinence Syndrome. This trial is designed to see if the use of sublingual (under the tongue) buprenorphine is able to be used safely and easily in newborns with the neonatal abstinence syndrome. Secondary goals will be to see if treatment with buprenorphine is associated shorter stays in the hospital and fewer days of treatment than the use of standard therapy. Another secondary goal will be to understand buprenorphine concentration in the blood of babies treated with the drug (this is called "pharmacokinetics").

ELIGIBILITY:
Inclusion Criteria:

* ≥ 37 weeks gestation
* exposure to opiates in utero
* demonstration of signs and symptoms of neonatal abstinence syndrome requiring treatment

Exclusion Criteria:

* major congenital malformations and/or intrauterine growth retardation
* medical illness requiring intensification of medical therapy
* concomitant benzodiazepine or severe alcohol abuse, self-report of regular use of alcohol or of benzodiazepines use in the past 30 days, and/or receipt of benzodiazepines by prescription (as determined by self-report or intake urine) by the mother during pregnancy,
* concomitant use of CYP 3A inhibitors (erythromycin, clarithromycin, ketoconazole, itraconazole, HIV protease inhibitors) or inducers (rifampin, carbamazepine, phenobarbital) prior to initiation of NAS treatment
* seizure activity or other neurologic abnormality
* breast feeding
* inability of mother to give informed consent due to co-morbid psychiatric diagnosis
* hypoglycemia requiring treatment with intravenous glucose

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Sublingual Buprenorphine safety and tolerability in the neonate | Index hospitalization

SECONDARY OUTCOMES:
Buprenorphine Pharmacokinetics | Index hospitalization
Efficacy: Length of treatment | Index hospitalization
Efficacy: Length of hospitalization | Index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, MS, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Kraft WK, Gibson E, Dysart K, Damle VS, Larusso JL, Greenspan JS, Moody DE, Kaltenbach K, Ehrlich ME. Sublingual buprenorphine for treatment of neonatal abstinence syndrome: a randomized trial. Pediatrics. 2008 Sep;122(3):e601-7. doi: 10.1542/peds.2008-0571. Epub 2008 Aug 11. PMID 18694901
- [Result] Kraft WK, Dysart K, Greenspan JS, Gibson E, Kaltenbach K, Ehrlich ME. Revised dose schema of sublingual buprenorphine in the treatment of the neonatal opioid abstinence syndrome. Addiction. 2011 Mar;106(3):574-80. doi: 10.1111/j.1360-0443.2010.03170.x. Epub 2010 Oct 6. PMID 20925688